CLINICAL TRIAL: NCT00520455
Title: Randomized Controlled Trial of Advanced Provision Emergency Contraception Among Women With Gonorrhea or Chlamydia
Brief Title: Randomized Trial of Advanced Provision Emergency Contraception Among Women With Gonorrhea or Chlamydia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 037249C
Record Dates: First submitted 2007-08-22; First posted 2007-08-24 (Estimated); Last update posted 2007-11-15 (Estimated); Status verified 2007-11

CONDITIONS: Pregnancy
MeSH Terms: interventions — Levonorgestrel; Condoms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): Control participants were advised where they could obtain hormonal contraception on a sliding scale basis. Participants were also advised where they could obtain hormonal contraception on a sliding scale basis.
- Intervention (Experimental): Study subjects were prescribed levonorgestrel 0.75mg taken twice 12 hours apart (Plan B) and a package of 30 condoms provided via a commerical pharmacy at no cost to the study subject. The subject could refill this prescription as many times as they wanted for 12 months
  Interventions: Drug: levonorgestrel 0.75mg taken twice 12 hours apart (Plan B) and condoms

INTERVENTIONS:
Drug: levonorgestrel 0.75mg taken twice 12 hours apart (Plan B) and condoms — levonorgestrel 0.75mg taken twice 12 hours apart (Plan B). Study subjects to take medication after unprotected vaginal intercourse
  Other Names: Plan B
  Arms: Intervention

SUMMARY:
The purpose of this trial is to determine whether providing non-contracepting women with gonorrhea or chlamydial infection with advanced provision emergency contraception (APEC) and condoms decreases their risk of becoming pregnant.

ELIGIBILITY:
Inclusion Criteria:

Non-contracepting women >15 years of age who were reported to Public Health Seattle & King County with a diagnosis for gonorrhea or chlamydial infection and who were interviewed by public health staff for purposes of partner notification

Exclusion Criteria:

* Use of effective contraception (hormonal contraception, IUD, diaphragm); sex with only one partner in the preceding 60 days who was status post vasectomy; age <15; inability to speak English; history of tubal ligation, hysterectomy, or menopause.

Ages: 16 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 177 (Actual)
Dates: Start 2004-01; Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
Pregnancy | 1 year - measured via interview every 3 months

SECONDARY OUTCOMES:
Abortion | 1 year - measured via interview every 3 months
Condom use | Measured every 3 months for one year
Use of hormonal contraception | Measured via interview every 3 months for one year

CONTACTS AND LOCATIONS:
Overall Officials: Matthew R Golden, MD, MPH, Principal Investigator — University of Washington
Locations (1):
- Public Health - Seattle & King County STD Clinic, Seattle, Washington, United States